CLINICAL TRIAL: NCT03706404
Title: Randomised Controlled Trial to Assess a Renal Colic Fast Track Pathway in the Emergency Department Using Point-of-care Ultrasound and Point-of-care Testing.
Brief Title: Renal Colic Fast Track Pathway in the Emergency Department.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Yale Tung Chen, Attending physician, Fellow director of the ultrasound division in the emergency department, principal investigator., Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: URGG/HULP_2018_03
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Renal Colic
Keywords: Renal Colic; Point-of-Care ultrasound; Point-of-Care testing
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care Testing and Ultrasound pathway (Experimental)
  Interventions: Diagnostic Test: Point-of-Care ultrasound and testing
- Classical pathway (No Intervention)

INTERVENTIONS:
Diagnostic Test: Point-of-Care ultrasound and testing — Point-of-Care ultrasound + Point-of-Care blood gas testing
  Arms: Point-of-care Testing and Ultrasound pathway

SUMMARY:
Validation of a high-resolution, fast track pathway that combines the use of laboratory tests at the Point-of-Care Testing (POCT) and Point-of-Care ultrasound (POCUS) versus the classical pathway, in which blood samples are sent to the central laboratory and comprehensive radiological exams ordered, being equally effective, at a lower cost of care and time of stay in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* First renal colic episode
* Need of analgesia
* Oral tolerance

Exclusion Criteria:

* Hemodynamic instability
* Fever
* Anuria
* Abdominal trauma
* Chronic renal failure
* Active oncologic disease
* Kidney transplant or monorenal patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Length of stay in the Emergency Department | 24 hours
Adverse events | 30 days

SECONDARY OUTCOMES:
Number of conclusive exams in the Point-of-Care intervention arm. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tung Chen Y, Rodriguez Fuertes P, Oliver Saez P, Villen Villegas T, Buno Soto A, Fernandez Calle P, Carballo Cardona C, Cobo Mora J, Jaen Canadas M, Yan Tong H, M Borobia A. Efficacy of a fast-track pathway for managing uncomplicated renal or ureteral colic in a hospital emergency department: the STONE randomized clinical trial of Sonography and Testing of a Nephrolithiasis Episode. Emergencias. 2021 Feb;33(1):23-28. English, Spanish. PMID 33496396